CLINICAL TRIAL: NCT04127006
Title: Rate of Progression in EYS Related Retinal Degeneration (Pro-EYS)
Brief Title: Rate of Progression in EYS Related Retinal Degeneration
Acronym: Pro-EYS
Status: Active, not recruiting | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Foundation Fighting Blindness (Other)
Responsible Party: Sponsor
Other Study IDs: Pro-EYS
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Retinitis Pigmentosa; Eye Diseases
Keywords: EYS mutation; Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa; Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vision Cohort 1: Participants with the better eye Screening Visit visual acuity ETDRS letter score of 54 or more [approximate Snellen equivalent 20/80 or better] and visual field diameter 10 degrees or more in every meridian of the central field
- Vision Cohort 2: Participants with the better eye Screening Visit visual acuity ETDRS letter score of 19-53 [approximate Snellen equivalent 20/100 - 20/400] or (visual acuity ETDRS letter score of 54 or more [approximate Snellen equivalent 20/80 or better] and visual field diameter less than 10 degrees in any meridian of the central field)
- Vision Cohort 3: Participants with the better eye Screening Visit visual acuity ETDRS letter score of 18 or less [approximate Snellen equivalent 20/500 or worse]

SUMMARY:
The overall goal of this project funded by the Foundation Fighting Blindness is to characterize the natural history of disease progression in patients with EYS mutations in order to accelerate the development of outcome measures for clinical trials.

DETAILED DESCRIPTION:
This natural history study of patients with EYS mutations will accelerate the development of outcome measures for clinical trials. Sensitive, reliable outcome measures of retinal degeneration will greatly facilitate development of treatments for retinitis pigmentosa due to EYS mutations. Together these approaches are expected to have an impact on understanding EYS-related retinal degeneration, developing experimental treatment protocols, and assessing their effectiveness.

The goals and expected impact of this natural history study are to:

1. Describe the natural history of retinal degeneration in patients with biallelic mutations in the EYS gene
2. Identify sensitive structural and functional outcome measures to use for future multicenter clinical trials in EYS-related retinal degeneration
3. Identify well-defined subpopulations for future clinical trials of investigative treatments for EYS-related retinal degeneration

Study Objectives

The primary objectives of the natural history study are to:

1. Characterize the natural history of retinal degeneration associated with biallelic pathogenic mutations in the EYS gene over 4 years, as measured using functional, structural, and patient-reported outcome measures
2. Investigate whether structural outcome measures can be validated as surrogates for functional outcomes in individuals with biallelic pathogenic mutations in the EYS gene
3. Evaluate possible risk factors (genotype, phenotype, environmental, and comorbidities) for progression of the outcome measures at 4 years in individual with biallelic pathogenic mutations in the EYS gene
4. Evaluate variability and symmetry of left and right eye outcomes over 4 years in individuals with biallelic pathogenic mutations in the EYS gene

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study and able to communicate consent during the consent process
2. Ability to return for all study visits over 48 months
3. Age ≥ 18 years
4. Must meet one of the Genetic Screening Criteria, defined below:

   * Screening Group A: At least 2 disease-causing variants in the EYS gene which are homozygous or heterozygous in trans, based on a report from a clinically-certified lab (or a report from a research lab that has been pre- approved by the Genetics Committee)
   * Screening Group B: Only 1 disease-causing variant in the EYS gene, based on a report from a clinically-certified lab (or a report from a research lab which has been pre-approved by the Genetics Committee)
   * Screening Group C: At least 2 disease-causing variants in the EYS gene which are unknown phase, based on a report from a clinically-certified lab (or a report from a research lab which has been pre-approved by the Genetics Committee)

Note pertaining to all Screening Groups: if a participant has a variant(s) of unknown significance, he/she would still qualify as long as there is at least 1 disease-causing variant(s) on the EYS gene.

Ocular Inclusion Criteria:

Both eyes must meet all of the following:

1. Clinical diagnosis of retinal dystrophy
2. Clear ocular media and adequate pupil dilation to permit good quality photographic imaging

Exclusion Criteria:

1. Mutations in genes that cause autosomal dominant retinitis pigmentosa (ADRP), X-linked retinitis pigmentosa (RP), or presence of biallelic mutations in autosomal recessive RP/retinal dystrophy genes other than EYS
2. Expected to enter experimental treatment trial at any time during this study
3. History of more than 1 year of cumulative treatment, at any time, with an agent associated with pigmentary retinopathy (including hydroxychloroquine, chloroquine, thioridazine, and deferoxamine)

Ocular exclusion Criteria:

If either eye has any of the following, the participant is not eligible:

1. Current vitreous hemorrhage
2. Current or any history of rhegmatogenous retinal detachment
3. Current or any history of (e.g., prior to cataract or refractive surgery) spherical equivalent of the refractive error worse than -8 Diopters of myopia
4. History of intraocular surgery (e.g., cataract surgery, vitrectomy, penetrating keratoplasty, or LASIK) within the last 3 months
5. Current or any history of confirmed diagnosis of glaucoma (e.g., based on glaucomatous VF changes or nerve changes, or history of glaucoma filtering surgery)
6. Current or any history of retinal vascular occlusion or proliferative diabetic retinopathy
7. History or current evidence of ocular disease that, in the opinion of the investigator, may confound assessment of visual function
8. History or evidence of active treatment for retinitis pigmentosa that could affect the progression of retinal degeneration, including:

   1. Any use of ocular stem cell or gene therapy
   2. Any treatment with ocriplasmin
   3. Treatment with an ophthalmic oligonucleotide within the last 9 months (last treatment date is less than 9 months prior to Screening Visit date)
   4. Treatment with any other product within five times the expected half-life of the product (time from last treatment date to Screening Visit date is at least 5 times the half-life of the given product)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential eligibility may be assessed as part of a routine care examination by an investigator prior to obtaining informed consent, as part of usual care, by referral from another physician, or self-referral.
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Field Sensitivity | Baseline and every year until study completion (4 years)
  Measured by static perimetry with topographic analysis (Hill of Vision) and assessed by a central reading center for cohorts 1 and 2.
Change in Best Corrected Visual Acuity | Screening visit and every year until study completion (4 years) with the exception of baseline for cohorts 1 and 2. Screening visit and 48 month follow-up for cohort 3.
  Measured on the Electronic Visual Acuity (EVA) system or ETDRS charts. Berkeley Rudimentary Vision Test (BRVT) will be used for patients unable to see letters.
Change in Mean Retinal Sensitivity | Baseline and every year until study completion (4 years).
  Measured by fundus-guided microperimetry (MP) and assessed by a central reading center at selected sites with requisite equipment for cohorts 1 and 2.
Change in Full-field Retinal Sensitivity | Baseline and every year until study completion (4 years) for cohort 1 and 2. Baseline and 4 year follow-up for cohort 3.
  Measured by full-field stimulus threshold (FST) testing to blue, white, and red stimuli
Change in Best Corrected Low Luminance visual acuity | Screening visit and every year until study completion (4 years) with the exception of baseline for cohorts 1 and 2. Screening visit and 48 month follow-up for cohort 3.
  Measured by letter score
Change in Contrast Sensitivity Function | Baseline and every year until study completion (4 years).
  Measured by the CSV-1000E VectorVision chart for cohorts 1 and 2.
Change in Retinal Function | Baseline and 4 year follow-up visit.
  Measured by full-field electroretinogram (ERG) amplitudes and timing in response to rod- and cone-specific stimuli for cohorts 1 and 2.
Change in Ellipsoid zone (EZ) area | Baseline and every year until study completion (4 years) for cohorts 1 and 2. Baseline and 4 year follow-up for cohort 3.
  Measured by spectral domain optical coherence tomography (SD-OCT) and assessed by a central reading center

SECONDARY OUTCOMES:
Explore Qualitative categorization of Fundus Autofluorescence (FAF) pattern | Baseline and every year until study completion (4 years) for cohorts 1 and 2. Baseline and 4 year follow-up for cohort 3.
  Assessed by a central reading center
Explore quantitative measures of FAF | Baseline and every year until study completion (4 years) for cohorts 1 and 2. Baseline and 4 year follow-up for cohort 3.
  assessed by a central reading center

OTHER OUTCOMES:
Patient Reported Outcomes for Vision Cohorts 1 and 2 (Vision Visual Functioning) | Baseline, 2 year follow-up, and 4 year follow-up visit
  Measured by Veterans Affairs Low Vision Visual Functioning Questionnaire (VA LV VFQ-48)
Patient Reported Outcomes for Vision Cohorts 1 and 2 | Baseline, 2 year follow-up, and 4 year follow-up visit
  Measured by Patient-Reported Outcomes Measurement Information System (PROMIS®-29)
Patient Reported Outcomes for Vision Cohort 3 (Vision Visual Functioning) | Baseline and 4 year follow-up visit
  Measured by Ultra-Low Vision Visual Functioning Questionnaire (ULV-VFQ-50)
Patient Reported Outcomes for Vision Cohort 3 | Baseline and 4 year follow-up visit
  Measured by Patient-Reported Outcomes Measurement Information System (PROMIS®-29)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pennesi, MD, PhD, Study Chair — Retina Foundation of the Southwest
Locations (19):
- United States (13):
  - University of California, San Francisco, San Francisco, California
  - Colorado Retina Associates, Denver, Colorado
  - Vitreo-Retinal Associates, Gainesville, Florida
  - University of Miami: Neuro-ophthalmology Department, Miami, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - Kellogg Eye Center, University of Michigan, Ann Arbor, Michigan
  - Duke University Eye Center, Durham, North Carolina
  - Oregon Health Science University Casey Eye Institute, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Retina Foundation of the Southwest, Dallas, Texas
  - University of Wisconsin-Madison: McPherson Eye Research Institute, Madison, Wisconsin
- Hospital for Sick Children, Toronto, Canada
- Helsinki University Hospital, Helsinki, Finland
- Centre hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris, France
- University of Tubingen, Tübingen, Germany
- Hadassah Medical Center, Jerusalem, Israel
- Radboud University, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
A de-identified database is placed in the public domain on the FFB/Jaeb public website after the completion of each protocol and publication of the manuscript.
Supporting Information: Study Protocol, ICF
Time Frame: After manuscript is published
Access Criteria: Users accessing data must enter an email address

REFERENCES:
- See also: Foundation Fighting Blindness Public Website — https://public.jaeb.org/ffb

DOCUMENTS (1):
  • Study Protocol (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT04127006/Prot_001.pdf